CLINICAL TRIAL: NCT00221611
Title: Intrathecal Administration of Baclofen (ITB) to Cerebral Palsy Patients With Therapy-Resistant Spasticity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1999/152
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Administration of intrathecal baclofen

SUMMARY:
Evaluation of the effect of intrathecal administration of Baclofen on spasticity of cerebral palsy patients, by means of standardized and internationally accepted scales

DETAILED DESCRIPTION:
Evaluation of the effect of intrathecal administration of Baclofen on spasticity of cerebral palsy patients, by means of standardized and internationally accepted scales

ELIGIBILITY:
Inclusion Criteria:

* CP patients with therapy-resistent spasticity
* Patients with sufficient body weight in relation to the volume
* Oral medication has failed: insufficient effect or too many side-effects
* The patient and family understand the objectives of the treatment and accept those objectives
* Informed Consent

Exclusion Criteria:

* Contra-indications for surgery (e.g. infection)
* Hypersensitivity to oral Baclofen

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80
Dates: Start 2000-01; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Spasticity of patients after 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Uyttendale, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be